CLINICAL TRIAL: NCT06489743
Title: Effect of Supplemental Oxygen Therapy (SOT) on 6-minute Walk Distance (6MWD) in Highlanders With High Altitude Pulmonary Hypertension Permanently Living at >2500m
Brief Title: Highlanders With High Altitude Pulmonary Hypertension (HAPH), 6 Minute Walk Distance (6MWD) Assessed at 3200m With and Without Supplemental Oxygen Therapy (SOT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HAPH_SOT_6MWT
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: High Altitude Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Hypoxia; High Altitude; Supplemental Oxygen Therapy; 6-Minute Walk Test
MeSH Terms: conditions — Pulmonary edema of mountaineers; Hypertension, Pulmonary; Hypoxia; Altitude Sickness

STUDY DESIGN:
Intervention Model Description: Each highlander with HAPH will perform a 6 MWT with and without SOT according to a cross-over design.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ambient air (Active Comparator): Highlanders with HAPH will perform the 6 MWT on ambient air at 3200 m
  Interventions: Other: 6-minute walk test (6MWT)
- SOT via nasal canula (Experimental): Portable pulsed supplemental oxygen therapy (SOT) will be provided via a nasal cannula from a regular portable oxygen concentrator carried on the back according to standard care
  Interventions: Other: 6-minute walk test (6MWT)

INTERVENTIONS:
Other: 6-minute walk test (6MWT) — 6-minute walk test (6MWT) will be performed according to clinical standards

SUMMARY:
The investigators aim to study the effect of SOT in highlanders with high altitude pulmonary hypertension (HAPH) who permanently live >2500m on 6-minute walk distance (6MWD) assessed at 3200m.

DETAILED DESCRIPTION:
Highlanders with HAPH diagnosed by echocardiography and defined by a RV/RA (Tricuspid Regurgitation Pressure Gradient) >30 mmHg will be recruited for this project. Highlanders permanently living at HA >2500 m will perform a 6-minute walk distance test near their living altitude in Aksay at 3200 m with and without portable pulsed supplemental oxygen therapy (SOT) via nasal cannula according to a randomized cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* Permanently living >2500 m
* HAPH diagnosed with a minimum RV/RA of 30 mmHg assessed by echocardiography at an altitude of 3200 m
* Written informed consent

Exclusion Criteria:

* Highlanders who cannot follow the study investigations,
* Patients with moderate to severe concomitant lung disease (FEV1<70% or forced vital capacity <70%), severe parenchymal lung disease, heavy smoking >20 cigarettes/day or >20 pack-years.
* Coexistent unstable systemic hypertension or coronary artery disease that required adjustment of medication within the last 2 months
* Regular use of medication that affects control of breathing (benzodiazepines, opioids, acetazolamide)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
6-minute walk distance (6MWD) with SOT vs. ambient air at 3200 m | after 6 minute
  Change in 6MWD in meters between SOT vs. ambient air at 3200 m

SECONDARY OUTCOMES:
SpO2 at rest and end 6MWT with SOT vs. ambient air at 3200 m | after 6 minute
  Change of the arterial oxygen saturation by pulse oximetry (SpO2) at rest and at end of the 6MWT with SOT vs. ambient air at 3200 m
Heart rate at rest and end 6MWT with SOT vs. ambient air at 3200 m | after 6 minute
  Change of the heart rate at rest and at end of the 6MWT with SOT vs. ambient air at 3200 m
Blood pressure at rest and end 6MWT with SOT vs. ambient air at 3200 m | after 6 minute
  Change of the blood pressure at rest and at end of the 6MWT with SOT vs. ambient air at 3200 m
Borg Dyspnea scale at end 6MWT with SOT vs. ambient air at 3200 m | after 6 minute
  Change of the Borg CR10 dyspnea scale at end of the 6MWT with SOT vs. ambient air at 3200 m
Borg leg fatigue scale at end 6MWT with SOT vs. ambient air at 3200 m | after 6 minute
  Change of the Borg CR10 leg fatigue scale at end of the 6MWT with SOT vs. ambient air at 3200 m

CONTACTS AND LOCATIONS:
Overall Officials: Talant MA Sooronbaev, Prof. Dr., Principal Investigator — National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov; Silvia Ulrich, Prof. Dr., Principal Investigator — University Hospital Zurich, Department of Pulmonology
Locations (1):
- Aksay Medical Center, Aksay Plateau, Naryn Region, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided